CLINICAL TRIAL: NCT03179098
Title: Immediate Effects of Superficial Heat Associated With Sustained Stretching on Post-traumatic Elbow Contracture: a Randomized Clinical Trial
Brief Title: Immediate Effects of Superficial Heat Associated With Elongation in the Posttraumatic Elbow Contracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marisa de Cassia Registro Fonseca, University of Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FMRPUSP2
Record Dates: First submitted 2017-01-29; First posted 2017-06-07 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Contracture of Elbow Joint
Keywords: Elbow; Stretching; Joint amplitude; Electromyography; Surface heat; Orthosis; Posttraumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (GC) (Active Comparator): The control group (GC) that will perform the 10 'sustained stretching tractioned by a load proportional to the force captured during a maximal voluntary isometric contraction (MVIC)
  Interventions: Other: CIVM; Other: GC- Sustained Stretching
- GWM (Active Comparator): The modified Weeks Group (GWM) that will carry out the modified Weeks protocol
  Interventions: Other: Modified Weeks protocol; Other: CIVM

INTERVENTIONS:
Other: Modified Weeks protocol — The modified Weeks group (GWM) will apply the protocol suggested by Flowers (2002), the positioning will be maintained and at rest will be done electromyographic registers, active goniometry and EVA. Soon afterwards the patients will be submitted to the whirlwind for 20 minutes at a temperature of 41 ° C performing active flexion and elbow extension movements. After the swirl the patients will be submitted to a stretching maintained for 10 minutes with load proportional to the force captured during MVIC according to the pain of the patient. The load will be positioned through a leather device 20 cm from the lateral epicondyle of the elbow.
  Arms: GWM
Other: CIVM — Patients underwent electromyographic analysis for the determination of maximal voluntary isometric contraction. The force will be collected for 5 seconds during a CIVM, in which a load cell model MM50 (Kratos, Cotia, SP, Brazil) will be positioned between the floor and the forearm of the volunteer, being coupled to a leather device at 20 cm Make the lateral epicondyle of the elbow. The angle between the forearm and the cable containing a load cell with a 90 degree service.
Other: GC- Sustained Stretching — The control group will be applied to sustained stretching, patients will be placed in the supine position with abduction of the shoulder of 30 ° in the plane of the scapula and the forearm in neutral throughout the entire test and the elbow will be supported in a towel to avoid discomfort And compression in the region of the olecranon.
  Arms: Control group (GC)

SUMMARY:
The elbow contracture is a secondary injury that can occur after direct trauma, causing the patient to have limitations in their range of motion. Objective evaluation protocols that help in decision making for the indication of these therapeutic resources have great value in rehabilitation, as they reduce unnecessary expenses and improve the assertiveness in the indication of this resource.

Objective: To verify the immediate effects of superficial heat associated with sustained stretching through muscle activity and range of motion in the posttraumatic contractures of the elbow seeking the best indication of orthosis.

Methods: Characterized as a randomized crossover type clinical trial. Sample of 20 adult subjects, of both sexes, over 18 years old, with elbow stiffness due to fractures and / or dislocations with indication of orthosis use. Patients will be divided into 2 randomly assigned intervention groups: the control group (CG) who will perform the 10 'sustained stretching drawn by a defined load through maximal voluntary isometric contraction (MVIC) and the modified Weeks Group (GWM) will perform 20 'of surface heat through the swirl and soon after the stretching sustained by 10' with already defined load. All patients will undergo an initial assessment and will participate in all 2 interventions while respecting a 7 day washout period. Goniometry and the visual analogue scale will be applied at the beginning and end of the interventions. The Delsys® brand equipment will be used to collect the electromyographic data. Placement and positioning of the electrodes will follow the determinations of the Seniam protocol. The activation of the brachial, brachioradial and triceps brachii muscles during the MVIC will be analyzed and also during the respective intervention protocols.

ELIGIBILITY:
Inclusion:

* patients between the ages of 18 and 60
* of both sexes
* who present elbow stiffness with flexural contractures resulting from fractures and / or dislocations,
* who are in the stages of fibroblastic healing and remodeling
* will be selected, with indication of use of bracing for gain of range of motion
* whether or not undergoing rehabilitation either after conservative or surgical orthopedic treatment

Exclusion:

* Individuals who have clinical or surgical restrictions to perform activities of daily living
* therapeutic exercises or use of orthoses
* who have lesions in the central nervous system
* open lesions
* moderate to high intensity pain to sustained passive stretching

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Range of motion of elboww | 10 minutes
  Goniometry of maximal elbow extension (degrees)

SECONDARY OUTCOMES:
Surface electromyography | 10 minutes
  Electromyographic activity of the agonist and elbow antagonist muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Lucy Montoro Institute of Rehabilitation, Ribeirão Preto, São Paulo, Brazil